CLINICAL TRIAL: NCT06252389
Title: Treating Achilles Tendon Rupture Complicated by Pre-existing Tendinopathy With Repair Augmented With a Bioinductive Collagen Implant
Brief Title: Degenerative Achilles Tendon Rupture Repair With Regeneten Augmentation
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: AchillesRegeneten
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Achilles Tendon Rupture; Achilles Tendinopathy
Keywords: Achilles; Regeneten; Tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Achilles Regeneten: bovine collagen patch to augmented repair in acute Achilles tendon rupture with pre-existing tendinopathy
  Interventions: Procedure: Achilles Tendon Repair augmented with Bioinductive Collagen Patch

INTERVENTIONS:
Procedure: Achilles Tendon Repair augmented with Bioinductive Collagen Patch — Standard Achilles Tendon Repair augmented with Bioinductive Collagen Patch. Standard Rehabilitation Protocol.

SUMMARY:
Retrospective Case Series to investigate the effect a bovine collagen patch to augmented repair in acute Achilles tendon rupture with pre-existing tendinopathy

DETAILED DESCRIPTION:
Retrospective Case Series. Investigate the effect a bovine collagen patch to augmented repair in acute Achilles tendon rupture with pre-existing tendinopathy.

Acute Achilles tendon rupture patients all underwent pre-operative ultrasound; those with tendinopathy enrolled into study.

Standard Achilles tendon repair performed; augmented with a bioinductive collagen patch (Regeneten)

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative ultrasound confirmation of tendinopathy

Exclusion Criteria:

* Underwent lower limb intervention with past 3 months
* Physical or psychological condition impairing ability to consent
* Physical or psychological condition impairing ability to adhere to rehabilitation protocol
* allergy to bovine material
* pregnant individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals admitted with an acute Achilles tendon rupture
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Outcome Score (FAOS) | 2 weeks, 6 weeks, 3 months, 6 months
  Symptoms measured by the patient reported outcome measure FAOS. It is split into 5 sections including: Symptoms, Pain, ADL function, Sporting activity, and Quality of Life.

SECONDARY OUTCOMES:
Victoria Institute of Sports Assessment - Achilles (VISA-A) | 2 weeks, 6 weeks, 3 months, 6 months
  Symptoms measured by the Achilles specific patient reported outcome measure VISA-A.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: No